CLINICAL TRIAL: NCT06050889
Title: Mechanisms of Exercise-Induced Hypoalgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Abigail Wilson, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Exercise (Experimental): Participants will complete an upper body resistance exercise until they report a high fatigue level.
  Interventions: Other: Positive Expectations Instructional Set; Other: Negative Expectations Instructional Set
- Low Intensity Exercise (Experimental): Participants will complete an upper body resistance exercise until they report a low fatigue level.
  Interventions: Other: Positive Expectations Instructional Set; Other: Negative Expectations Instructional Set

INTERVENTIONS:
Other: Positive Expectations Instructional Set — Participants randomly assigned to this instructional set will be told, "You will be completing an intervention known to be effective for some people with shoulder pain. We expect this will make you less sensitive to the pressure applied to your shoulder and thigh and you will require more pressure than what was previously necessary to experience pain."
Other: Negative Expectations Instructional Set — Participants randomly assigned to this instructional set will be told, "You will be completing an intervention which is not effective for some people with shoulder pain. We expect this will make you more sensitive to the pressure applied to your shoulder and thigh and you will require less pressure than what was previously necessary to experience pain."

SUMMARY:
Exercise-Induced Hypoalgesia (EIH) is a lessening of pain sensitivity in response to an acute bout of exercise. Limited research has examined the effects of expectations on EIH during a dynamic resistance training during different intensities. Therefore, the purpose of this study is to examine the effects of positive and negative expectations on EIH.

DETAILED DESCRIPTION:
Individuals who meet the eligibility criteria and consent to participate will attend one testing session that is approximately one hour. Baseline Pressure Pain Threshold will be measured followed by random assignment to one of four study arms.

ELIGIBILITY:
Inclusion Criteria:

* Pain Free

Exclusion Criteria:

* Non-English speaking
* Regular use of prescription pain medications
* Current or history of chronic pain condition
* Currently taking blood-thinning medication
* Any blood clotting disorder, such as hemophilia
* Systemic medical condition known to affect sensation, such as uncontrolled diabetes or neurological conditions
* Not physically ready to exercise without a medical exam as indicated by the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Not have had Surgery, injury, or fracture within the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | Change from baseline immediately after exercise
  Pressure Pain Threshold will be applied with a digital algometer before and after the exercise intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States